CLINICAL TRIAL: NCT04073563
Title: Prospective, Randomized, Controlled, Blinded Pivotal Study In Subjects Undergoing A Transforaminal Lumbar Interbody Fusion (TLIF) At One Or Two Levels Using Infuse™ Bone Graft With an Intervertebral Body Fusion Device and Posterior Supplemental Fixation For The Treatment Of Symptomatic Degenerative Disease Of The Lumbosacral Spine
Brief Title: Transforaminal Lumbar Interbody Fusion (TLIF)
Acronym: TLIF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MDT17074SD1706
Record Dates: First submitted 2019-08-27; First posted 2019-08-29 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Degenerative Disease of the Lumbosacral Spine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Group #1 (Experimental): Investigational Infuse™ 2.1 mg/level with available local bone autograft and supplemented with cancellous allograft as needed
  Interventions: Device: Infuse™ Bone Graft (Infuse™); Device: Intervertebral body fusion device and Medtronic posterior Fixation Systems
- Group #2 (Experimental): Investigational Infuse™ 4.2 mg/level with available local bone autograft and supplemented with cancellous allograft as needed
  Interventions: Device: Infuse™ Bone Graft (Infuse™); Device: Intervertebral body fusion device and Medtronic posterior Fixation Systems
- Control (Active Comparator): Local bone autograft and supplemented with cancellous allograft as needed.
  Interventions: Device: Intervertebral body fusion device and Medtronic posterior Fixation Systems

INTERVENTIONS:
Device: Infuse™ Bone Graft (Infuse™) — (Recombinant human bone morphogenetic protein-2 (rhBMP-2)/absorbable collagen sponge (ACS))
  Arms: Group #1; Group #2
Device: Intervertebral body fusion device and Medtronic posterior Fixation Systems — Adaptix™Interbody System, Capstone™ Spinal System, Catalyft™ PL Interbody System

SUMMARY:
This is a global, multi-center, prospective, randomized, blinded, controlled pivotal study. Clinical and radiological evaluation will be performed preoperatively and postoperatively up to 24 months; and endpoint success will be determined at 24 months postoperatively.

Overall a maximum of 600 subjects will be enrolled and treated. The purpose of the study is to provide safety and effectiveness data of Infuse™ in Transforaminal Lumbar Interbody Fusion (TLIF) procedures and to obtain indication expansion for Infuse™ use in one and two level TLIF procedures.

ELIGIBILITY:
Inclusion Criteria:

A subject must meet all of the following inclusion criteria to participate in this study:

* I.1. Has degenerative disease of the lumbosacral spine in one or two adjacent levels (L2 to S1) that results in radiculopathy secondary to nerve root compression, manifested by:

  1. History of radiating leg or buttock pain, paresthesia, numbness or weakness, or
  2. History of neurogenic claudication.
* I.2. Has a history of low back pain.
* I.3. Has radiographic evidence (e.g. CT, MRI, x-ray, etc.) of degenerative lumbosacral disease including at least one of the following:

  1. Instability up to and including Grade 2 spondylolisthesis/retrolisthesis based on the Meyerding classification (Meyerding, HW, 1932), or lateral listhesis demonstrated by coronal plane translation (slippage) of the superior (cranial) vertebral body lateral to the inferior (caudal) vertebral body less than or equal to 3mm, or
  2. Stenosis, or narrowing, of the lumbar spinal canal and/or intervertebral foramen requiring significant decompression leading to segmental instability, or
  3. Recurrent disc herniation
* I.4. Has preoperative Oswestry Disability Index score ≥ 35.

Has to meet either inclusion criteria 5 or 6 to qualify for the study:

* I.5. Has preoperative back and leg pain scores of (back pain ≥ 4 and leg pain ≥ 1) based on the Preoperative Back and Leg Pain Questionnaire.
* I.6. Has preoperative back and leg pain scores of (back pain ≥ 1 and leg pain ≥ 4) based on the Preoperative Back and Leg Pain Questionnaire.
* I.7. Is at least 18 years of age and skeletally mature at the time of surgery.
* I.8. Has not responded to non-operative treatment (e.g., bed rest, physical therapy, medications, spinal injections, manipulation, and/or TENS) for a period of six months.
* I.9. Is willing and able to comply with the study plan and able to understand and sign the subject Informed Consent Form.

Exclusion Criteria:

A subject will be excluded from participating in this study for any of the following reasons:

* E.1 Prior surgical procedure at the involved or adjacent spinal levels (e.g. fusion, arthroplasty, and/or other non-fusion procedures). Prior discectomy and/or laminectomy at the target or adjacent levels is allowed.
* E.2 Significant lumbar instability defined as sagittal listhesis greater than Grade 2 at any involved level using the Meyerding Classification or lateral listhesis greater than 3 mm at any involved level.
* E.3 Planned use of an internal or external bone growth stimulator.
* E.4 Lumbar scoliosis >30 degrees.
* E.5 Patients who had a previous diagnosis of osteoporosis with a T-score of -2.5 or below in the last 12 months existing together with a prevalent fragility fracture. (If subject has a prevalent fragility fracture and a T-score hasn't been assessed in the last 12 months, a DEXA will need to be obtained.)
* E.6 Morbidly obese, as defined by a Body Mass Index (BMI) >40.
* E.7 Presence of active malignancy or prior history of malignancy (non-invasive basal cell carcinoma of the skin and non-invasive squamous cell carcinoma localized only to the skin is allowed).
* E.8 Overt or active bacterial infection, either local to surgical space or systemic.
* E.9 Has undergone administration of any type of corticosteroid, antineoplastic, immunostimulating, or immunosuppressive agents, or medications known to inhibit the healing of bone or soft tissue within 30 days prior to implantation of the assigned treatment.

  * This includes patients ≥ 65 years of age taking warfarin with documented diagnosed osteoporosis. All other patients taking warfarin should washout for at least 5 days prior to treatment
  * Use of steroidal inhalers is allowed pre- and post-operatively
  * Short-term steroidal use (e.g., Medrol Dosepak) is allowed pre and post-operatively. For this clinical study, short-term use is defined as ≤ two weeks. Use of steroids for longer than two weeks post-operatively through the 24-month follow-up visit is prohibited.
* E.10 Co-morbidities, which in the investigator's opinion, precludes the subject from being a surgical candidate.
* E.11 Autoimmune disease, which in the investigator's opinion, is known to affect bone metabolism or the spine (e.g., spondyloarthropathies, juvenile arthritis, rheumatoid arthritis, Graves' disease, Hashimoto's thyroiditis).
* E.12 Any endocrine or metabolic disorder, which in the investigator's opinion, is known to affect osteogenesis (e.g., Paget's disease, renal osteodystrophy, Ehlers-Danlos syndrome, or osteogenesis imperfecta).
* E.13 Known exposure to any recombinant proteins used for bone formation (e.g., Infuse™ Bone Graft, OP-1 Putty, OP-1 Implant, AUGMENT Bone Graft, GEM21S, i-FACTOR Peptide Enhanced Bone Graft, or PepGen P-15 Synthetic Bone Graft).
* E.14 Known hypersensitivity or allergy to any components of the study treatments including, but not limited to bone morphogenetic proteins (BMPs); injectable collagen; protein pharmaceuticals (e.g.,monoclonal antibodies or gamma globulins); bovine collagen products; and/or instrumentation materials (e.g., titanium, titanium alloy, cobalt chrome, cobalt chrome alloy, or PEEK).
* E.15 History of any allergy resulting in anaphylaxis.
* E.16 Is a prisoner.
* E.17 Is mentally incompetent. If questionable, obtain psychiatric consult.
* E.18 Treatment with an investigational therapy (drug, device, and/or biologic) targeting spinal conditions within 3 months prior to implantation surgery, treatment with any other investigational therapies within 30 days prior to implantation surgery, or such treatment is planned during the 24-month period following implantation of the study treatment.
* E.19 Pregnant or nursing. Females of child-bearing potential must agree not to become pregnant for 24 months following surgery.
* E.20 A documented diagnosis of substance use disorder as defined by the DSM-5.22 (Nicotine use is allowed.)
* E.21 Pursuing worker's compensation or active litigation for spinal fusion procedure.
* E.22 Any condition, which in the investigator's opinion, would interfere with the subject's ability to comply with study instructions, which might confound data interpretation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2019-12-19 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Overall success at 24 months | 24 months
  Overall success is defined as the participant who meet the following five criteria:
  * Pain/disability (ODI) success, defined as at least a 15-point improvement from baseline;
  * Fusion success as defined in primary outcome 2.
  * Neurological success, defined as maintenance or improvement in neurological status;
  * No SAE related to the TLIF grafting material or interbody device; and
  * No secondary surgeries at index level that are related to the TLIF grafting material or interbody device
Fusion success at 24 months | 24 Months
  Fusion success at each treatment level must demonstrate:
  * Evidence of bridging bone via CT. Solid fusion is based on evidence of continuous bone bridging from the superior to the inferior vertebral body at the target level(s) in at least 1 of the following locations: right lateral, left lateral, anterior, posterior, or through the intervertebral body fusion device.
  * No evidence of motion as defined by less than 2 mm translational motion and less than 3° in angular motion at each treated level (flexion/extension radiographs).

SECONDARY OUTCOMES:
Time to fusion | From surgery to 24 Months
  The first time point when a subject's fusion status has been determined to be a success per the fusion success criteria
ODI success | 24 months
  The self-administered Oswestry Disability Index (ODI) will be used. The ODI scale ranges from 0-100. The best score is 0 (no disability) and worst is 100 (maximum disability). Success will be defined as pain/disability improvement postoperatively according to the following definition: Preoperative Score - Postoperative Score ≥ 15 points
Leg pain success | 24 months
  Numerical rating scales (NRS 0-10) will be used to measure leg pain, with a score of 0 representing "no pain" and a score of 10 representing "pain as bad as it could be. Success for leg pain is defined as at least 30% improvement from pre-operative score: (Preoperative Score - Postoperative Score) / Preoperative Score ≥ 30%
Back pain success | 24 months
  Numerical rating scales (NRS 0-10) will be used to measure back pain, with a score of 0 representing "no pain" and a score of 10 representing "pain as bad as it could be". Success for back pain is defined as at least 30% improvement from pre-operative score: (Preoperative Score - Postoperative Score) / Preoperative Score ≥ 30%
Neurological success | 24 months
  Overall neurological success is defined as maintenance or improvement in four key neurological assessments: motor function, sensory function, reflexes, and straight leg raise. In order to be considered a success, each element in the motor, sensory, reflexes, and straight leg raise examinations must remain the same or improve from the time of the preoperative evaluation to the time period evaluated. Therefore, if any one motor, sensory, or reflexes element does not stay the same or improve, then a subject will not be considered a success for neurological status.
Serious Adverse Events | up to 24 months
  Serious Adverse Events related to TLIF grafting material or interbody device up to 24 months
Secondary Surgery | up to 24 months
  Secondary surgeries that are classified as a "failure", defined as any secondary surgeries at index level(s) "related" to TLIF grafting material or interbody device.

CONTACTS AND LOCATIONS:
Locations (46):
- United States (43):
  - Mayo Clinic, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - University of California Irvine, Irvine, California
  - Memorial Health Services, Laguna Hills, California
  - Cedars Sinai Spine Center, Los Angeles, California
  - University of California Davis Medical Center, Sacramento, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Boulder Neurosurgical Associates and Justin Parker Neurological Institute/E. Lee Nelson, Boulder, Colorado
  - Vail-Summit Orthopaedics and Neurosurgery, Vail, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Advent Health Altamonte Springs, Altamonte Springs, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Advent Health Orlando, Orlando, Florida
  - Orlando Health, Orlando, Florida
  - Foundation for Orthopaedic Research and Education, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Goodman Campbell Brain and Spine, Carmel, Indiana
  - Indiana Spine Group, Carmel, Indiana
  - OrthoIndy Northwest Office, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinic, Iowa City, Iowa
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Hospital for Special Surgery, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Mayfield Brain and Spine Clinic, Cincinnati, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Penn State-Hershey, Hershey, Pennsylvania
  - Rothman Institute, Philadelphia, Pennsylvania
  - Semmes Murphey, Memphis, Tennessee
  - Saint Thomas for Specialty Surgery, Nashville, Tennessee
  - Tennessee Orthopaedic Alliance, Nashville, Tennessee
  - DFW Center for Spinal Disorder, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - American Neurospine Institute, Plano, Texas
  - University of Virginia - Clinical Trial Office, Charlottesville, Virginia
  - University of Virginia - Health System, Charlottesville, Virginia
  - Swedish Neuroscience, Seattle, Washington
  - West Virginia University, 1 Medical Center Drive, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- China (3):
  - Peking University Third Hospital, Beijing
  - West China Hospital of Sichuan University, Chengdu
  - Chongqing Xinqiao Hospital Second Affiliated Hospital of Army Medical University, Chongqing